CLINICAL TRIAL: NCT04141553
Title: Gradual Diltiazem Infusion as an Approach to Initial Rate Control in Atrial Fibrillation or Atrial Flutter With Rapid Ventricular Response in the Emergency Setting
Brief Title: Bolus vs IVP (Intravenous Push) Diltiazem for Atrial Fibrillation or Flutter
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mercy Health Muskegon (Other)
Responsible Party: Principal Investigator, Joseph Betcher, MD, Principal Investigator, Mercy Health Muskegon
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RATE2019
Record Dates: First submitted 2019-10-15; First posted 2019-10-28 (Actual); Last update posted 2019-10-28 (Actual); Status verified 2019-10

CONDITIONS: Atrial Fibrillation; Atrial Flutter; Rapid Ventricular Response
MeSH Terms: conditions — Atrial Fibrillation; Atrial Flutter | interventions — Diltiazem; Saline Solution

STUDY DESIGN:
Intervention Model Description: A parallel randomized blinded model. Eligible and consented participants will be randomized to diltiazem IV push or diltiazem slow bolus. Each will receive an opposite sham infusion of saline provided as IVP push or slow bolus t0 maintain the blind. All participants will receive 30 mg oral dose of diltiazem. Standard of care measures will be provided concurrently as per routine care of patients with atrial fibrillation or atrial flutter with rapid ventricular response
  Participants will be randomized in 15 blocks of 20 to ensure there are equal numbers of participants in each group for interim analyses. The randomization scheme will allow for 300 participants to account for issues, including dropouts.
Who Masked: Care Provider
Masking Description: Randomization will be managed by unblinded emergency department pharmacist. This individual will have knowledge of the assigned treatment group for each participant, knowing if diltiazem is provided as IV push or slow infusion. Unblinded pharmacist will also provide sham saline dose, opposite of assigned diltiazem treatment to maintain the blind to care providers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Diltiazem IV push (Active Comparator): In the standard IV push group, diltiazem will be administered at a dose of 0.25 mg/kg, to a max dose of 25 mg, over 2 minutes. At time 0, these participants will also receive 30 mg of immediate release oral diltiazem. After 15 minutes, if adequate rate control of <110 BPM has not been achieved, an additional dose 0.35 mg/kg to a max dose of 35 mg will be administered. In order to maintain the blind, the control group will also receive 50 mL of 0.9% NS IV over 20 minutes.
  Interventions: Drug: Diltiazem Injection
- Diltiazem IV Slow Infusion (Active Comparator): In the slow infusion group, 50 mg of diltiazem will be diluted in 50 mL of 0.9% NS and infused over 20 minutes. Similar the other group, these participants will also receive 30 mg of immediate release oral diltiazem. In order to maintain the blind, this slow infusion group will receive the equivalent volume of IV 0.9% NS over 2 minutes as a placebo.
  Interventions: Drug: Diltiazem Injection

INTERVENTIONS:
Drug: Diltiazem Injection — Randomization to one of to active comparator groups
  Other Names: diltiazem immediate release oral tablet; 0.9% saline

SUMMARY:
The administration of intravenous non-dihydropyridine calcium channel blockers such as diltiazem for patients presenting in atrial fibrillation with rapid ventricular response, without evidence of pre-excitation, are recommended first-line therapies by the American Heart Association.1 Hypotension warrants careful consideration in the treatment of atrial fibrillation with a rapid ventricular response. Hemodynamic stability is a continuum, however, and rate control is often vital, particularly in patients who are refractory to electrical cardioversion [or who have underlying conditions such that tachycardia is not well tolerated]. Diltiazem has been utilized in dosing such as 2.5 mg/min in those with decreased blood pressure and atrial fibrillation with elevated ventricular rate.2 Lim et al. in 2002 demonstrated the effectiveness of a slow infusion of diltiazem 2.5 mg/min to a maximum of 50 mg to control rate in supraventricular tachycardia.

The study of the slow infusion of diltiazem has been limited to supraventricular tachycardia. No literature exists evaluating the efficacy of such a gradual infusion in atrial fibrillation or atrial flutter, rhythms affecting 2.7 million to 6.1 million Americans.1,3 It can be reasoned that a gradual infusion of diltiazem will minimize side effects, predominantly hypotension, and perhaps even demonstrate efficacy in alleviating hypotension due to decreased stroke volume from excessive tachycardia. The proposed benefits of an infusion, as compared to a bolus, would allow for the termination of an infusion as soon as rate control is achieved thus limiting the potential for hypotension. With current evidence-based literature validating the superiority of non-dihydropyridine calcium channel blockers and questions surrounding present recommendations of weight based intravenous dosing, the authors suggest an inquiry into the utility of a gradual infusion of diltiazem for initial rate control in patients presenting with atrial fibrillation or flutter with or without hypotension related to excessive tachycardia.

This is a prospective, randomized, double blind investigation to compare the effectiveness of standard IV (intravenous) push diltiazem at 0.25 mg/kg (to a maximum of 25 mg) over 2 minutes, with a potential repeat dose of 0.35 mg/kg if the initial dose is not effective versus a slow infusion of 50 mg of IV diltiazem diluted in 50 mL of 0.9% normal saline (NS) administered over 20 minutes. The investigators anticipate the data to be collected over the course of 2-3 years. These methods of diltiazem administration are already accepted practices at our institution and are consistent with current approved product labeling and professional judgment based upon clinical experience, and therefore the investigators do not foresee any additional risk to patients enrolled in our proposed study. In either treatment group, should hypotension or other clinical evidence of poor systemic perfusion, no additional IV diltiazem, or additional administration of a diltiazem infusion will be administered. The primary outcome measured will be the efficacy of treatment as defined by the obtainment of a heart rate of <110 beats/minute within 30 minutes of drug administration. Secondary outcomes evaluated will include the need for additional medications to achieve rate control including the need for repeat diltiazem bolus at 0.35 mg/kg, electrical cardioversion, admission, allergic reactions, and side effects including, but not limited to, systolic blood pressure less than 90 mmHg or bradycardia with heart rate less than 60 bpm.

ELIGIBILITY:
Inclusion Criteria:

* Be 18 years and older,
* Present with atrial fibrillation or atrial flutter with a rapid ventricular response
* Have a 12-lead ECG (electrocardiogram) showing atrial fibrillation or atrial flutter with a rapid ventricular rate greater than 120 beats per minute.
* Able to provide consent for self, or have a legally authorized representative available to provide consent by proxy.
* Have a cardiac history not inclusive of the diagnoses listed under exclusion criteria.

Exclusion Criteria:

* Altered mental status as a direct result of hemodynamic instability
* Heart rate >220 beats per minute
* 2nd or 3rd degree atrioventricular block
* QRS (time for ventricular repolarization) >110 milliseconds
* Temperature >38 Celsius
* Acute STEMI (ST-Elevation Myocardial Infarction)
* Pulmonary edema
* Unstable angina
* Allergy to diltiazem
* Pregnancy
* Breastfeeding
* History of pre-excitation syndrome
* Decompensated heart failure
* Incarcerated persons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2019-12-01 (Estimated); Primary Completion 2021-12-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Resolution of arrhythmia | within 30 minutes of drug administration
  Efficacy of treatment as defined by the achievement of a heart rate of <110 beats/minute

SECONDARY OUTCOMES:
Use of additional medications to achieve rate control | within 30 minutes of diltiazem administration
  Percentage of patients who require medications other than diltiazem to achieve rate control.
Frequency of cardioversion | within 30 minutes of diltiazem administration
  Incidence of electrical cardioversion to achieve rate control
Frequency of hospital admission | within 24 hours of study related treatment in the Emergency Department.
  Percentage of enrolled patients who require hospital admission to achieve and maintain rate control
Identification of adverse events. | at the time of diltiazem administration and and immediately following the medication
  Characterization and frequency of adverse events
Occurrence of allergic reactions | at the time of diltiazem administration and and immediately following the medication
  Evaluate occurrence of allergic reactions

IPD SHARING:
Plan to Share IPD: No
Data will not be shared